CLINICAL TRIAL: NCT06115889
Title: Smart Taiko-Drum Playing for Older Adults With Cognitive Frailty for Improving Cognitive and Physical Functions: A Randomized Controlled Feasibility Study
Brief Title: Smart Taiko-Drum Playing for Older Adults With Cognitive Frailty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P0046219
Record Dates: First submitted 2023-09-28; First posted 2023-11-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Impairment; Frailty
Keywords: Cognitive frailty; Motor-Cognitive Training; Drumming
MeSH Terms: conditions — Cognitive Dysfunction; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Trained research assistants will collect the data blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Taiko Drumming Group (Experimental): Smart Taiko Drumming
  Interventions: Behavioral: Smart Taiko Drumming
- Usual Care Waitlist Control Group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Smart Taiko Drumming — Participants will play drumming with the developed Smart Taiko Drumming System for 30-45 minutes three times per week for 16 weeks, in addition to usual care.
  Arms: Smart Taiko Drumming Group

SUMMARY:
The objective of this randomised controlled feasibility trial is to evaluate the feasibility of the Smart Taiko Drum-playing intervention embedding the cognitive-motor dual-task training concept for older adults with cognitive frailty, and identify the preliminary efficacy of the intervention on cognitive and physical functions and frailty status.

DETAILED DESCRIPTION:
1. Study design:

   - Randomized Control Trial
2. Participants:

   - Community-dwelling older adults with cognitive frailty
3. Setting:

   - Community centres for seniors
4. Intervention

   * Playing Smart Taiko three times/weeks x 16 weeks for 30 - 45 minutes each session
   * A Smart Taiko Drumming system has been developed for older adults to play the drumming game with their preferred music genres.
5. Waitlist-control group

   - Will receive usual care
6. Health outcomes that will be assessed three times at baseline, during (8th week) and immediate post-intervention (16th week)

   * cognitive functions
   * physical functions
   * mental health
   * physical frailty status
   * body composition
7. Feasibility evaluation

   * recruitment
   * retention
   * satisfactory survey
   * compliance with the survey
   * safety
   * focus group intervention with participants

ELIGIBILITY:
Inclusion Criteria:

* with cognitive frailty
* without a diagnosis of a neurological or psychiatric condition that could affect cognitive function
* live independently or with partial assistance
* with pre-frailty

Exclusion Criteria:

* with a significant sensory or motor impairment that would preclude participation in the intervention
* are unable to understand or follow instructions due to language or hearing impairment
* have already been in another cognitive or physical intervention programme within the past three months
* are taking medications that could significantly affect cognitive or physical functions
* with any medical condition or treatment that would contraindicate participation in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Attrition rate | Through study completion, an average of 2 years
  Overall attrition rate-defined as the proportion of participants at defined study points who discontinued the intervention or were lost to follow-up (calculated as number of participants that withdraw (numerator)/number of participants randomised (denominator)).
Recruitment rate | Through study completion, an average of 2 years
  The Proportion of eligible people recruited (= proportion of people randomised/proportion of people eligible).
Satisfaction to the intervention | Through study completion, an average of 2 years
  Satisfaction questionnaire, including questions of "Does the game provide an engaging environment for training?", "Do you think the exercise intensity suits you?"
Intervention Completion Rate | Through study completion, an average of 2 years.
  Overall intervention completion rate -defined as the proportion of participants who completed the allocated intervention with a minimum of 80% attendance.
  Calculated as number of participants allocated to the intervention that completed the minimum attendance (numerator)/number of participants allocated to treatment (denominator).

SECONDARY OUTCOMES:
Safety concerns of the intervention | Through study completion, an average of 2 years.
  Any adverse events during the intervention period
Overall cognitive function | 6 months
  The Hong Kong version of the Montreal Cognitive Assessment with the possible score from 0 - 30, with a higher score indicates better cognition
Executive function | 6 months
  Frontal Assessment Battery Total score with the possible score from 0 - 18, higher scores indicating better performance
Memory | 6 months
  Fuld Object Memory Evaluation Total Storage score ranges from 0 -50, with a higher score indicate better memory.
Verbal fluency | 6 months
  Modified Verbal Fluency Test will be used to assess the verbal fluency, with no highest score. Higher score indicates better verbal fluency.
Mobility and Balance | 6 months
  Time Up and Go Test will be used. The test measures how long it takes to stand up, walk a distance of 10 feet, turn, walk back, and sit down again. Shorter time indicate better mobility and balance.
Handgrip strength | 6 months
  To be measured with a hand-held Jamar Hand Dynamometer
Functional capacity and endurance | 6 months
  Six-Minute-Walk-Test. The longer distance walked indicates better functional capacity and endurance.
Mental wellbeing | 6 months
  Hospital Anxiety and Depression Scale is a 14-item measure designed to assess anxiety and depression symptoms. The total score ranges from 0 - 42, with a higher score indicates poorer mental wellbeing.
Happiness | 6 months
  Subjective Happiness Scale will be used. The four items will be responded on 7-Likert scale. The total is the average score of the 4-items, ranges from 1 - 7. Higher score is more happy.
Loneliness | 6 months
  De Jong Gierveld Loneliness Scale will be used. In this 6-item scale, three statements are made about 'emotional loneliness' and three about 'social loneliness'. Total score ranged from 0-6, with a higher score means higher loneliness.
Frailty status | 6 months
  FRAIL scale with the possible score range from 0 - 5. Higher score refers to higher frailty.
Body composition - Body weight | 6 months
  Bioelectrical impedance analysis will be used for measuring body composition using the InBody S10, Korea except those with contradictions, such as wearing a pacemaker.
Body composition - Skeletal muscle mass | 6 months
  Bioelectrical impedance analysis will be used for measuring body composition using the InBody S10, Korea except those with contradictions, such as wearing a pacemaker.
Body composition - body mass index | 6 months
  Body weight in kg is divided by square of body height
Body composition - body fat mass | 6 months
  Bioelectrical impedance analysis will be used for measuring body composition using the InBody S10, Korea except those with contradictions, such as wearing a pacemaker.
Body composition - percent body fat. | 6 months
  InBody S10, Korea except those with contradictions, such as wearing a pacemaker.

OTHER OUTCOMES:
Heart rate | 6 months
  Will be monitored for evaluating the intervention process

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Sze Ki Cheung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No